CLINICAL TRIAL: NCT07379736
Title: Randomised-Controlled Trial of an Online Brief Advice Intervention for Heavy Cannabis Users (RECALIBRATE)
Brief Title: Online Brief Advice Intervention for Heavy Cannabis Users
Acronym: Recalibrate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REMAS: 49272
Record Dates: First submitted 2025-09-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Cannabis User
Keywords: Cannabis; Brief Intervention
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational video (Experimental): A short educational video on cannabis withdrawal and personalised feedback on the Cannabis Withdrawal Scale
  Interventions: Other: Educational video
- Relaxation video (Active Comparator): A relaxation video and mood questionnaire
  Interventions: Other: Relaxation video

INTERVENTIONS:
Other: Educational video — Short educational video on cannabis withdrawal and personalised feedback on the Cannabis Withdrawal Scale.
  Other Names: Learning video; Informational video
  Arms: Educational video
Other: Relaxation video — Relaxation video and mood questionnaire with personalised feedback
  Other Names: Mindfulness video; Meditation video; Peaceful video
  Arms: Relaxation video

SUMMARY:
This project will evaluate whether a brief online intervention focused on cannabis withdrawal can increase awareness and insight about cannabis use disorder among daily cannabis users. The study will employ a randomised controlled trial design comparing an intervention consisting of a short educational video on cannabis withdrawal and personalised feedback on the Cannabis Withdrawal Scale, against a control condition of a relaxation video and mood questionnaire.

The investigators will aim to recruit at least 100 daily cannabis users (minimum 25 days of cannabis use /month and minimum 3.5g cannabis/week [low-medium daily use]) through Prolific, an online research participant platform. Potential participants will complete a brief screening questionnaire (1 minute) to confirm that participants meet inclusion criteria, before randomisation. The experiment will last 10-15 minutes and will include baseline demographic and substance use measures, the intervention or control condition, and outcome measures.

The primary outcome will be cannabis use awareness and insight as measured by the Substance Use Awareness and Insight Scale (SAS). Secondary outcomes will include intention to change cannabis use. This study aims to determine whether a short online intervention can increase awareness about cannabis withdrawal among heavy users. If successful, subsequent studies will be designed to assess these outcomes over the longer-term.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Daily/near daily cannabis users (25+ days/month, min. 3.5g/week)
* Sufficiently fluent in English

Exclusion Criteria:

* Participant is prescribed medical cannabis by a healthcare professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Substance (cannabis) use awareness and insight scale (SAS) | Day 1
  Measured by the Substance Use Awareness and Insight Scale, designed to assess awareness in substance use disorder. Minimum value = 0, maximum value 70. Higher score = worse outcome, less insight and awareness.

SECONDARY OUTCOMES:
Intention to change cannabis use | Day 1
  This outcome measures participants' motivation and readiness to alter their cannabis consumption behaviours following the intervention. The Intention to Change Cannabis Use scale will be used which is adapted from Motivation to Stop Scale. Minimum score = 1, maximum score = 7. Higher score = better outcome, higher motivation to stop.

CONTACTS AND LOCATIONS:
Locations (1):
- Denmark Hill, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No